CLINICAL TRIAL: NCT07159048
Title: A Prospective, Multi-center, Randomized Controlled Clinical Trial to Evaluate the Safety, Efficacy and Immune Response of Multimodal Thermal Therapy in the Treatment of Malignant Liver Tumors
Brief Title: The Safety, Efficacy, and Immune Response of Multimodal Thermal Therapy in the Treatment of Malignant Liver Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Lichao Xu, Associate Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-308-4457
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma; Colorectal Cancer Liver Metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Tumor Thermal Therapy (Experimental): These patients will receive multimodal thermal therapy using multimodal tumor thermal therapy system.
  Interventions: Device: Multimodal Tumor Thermal Therapy System
- Single Thermal Ablation (Experimental): These patients will receive local ablation using the microwave ablation system or radiofrequency ablation system.
  Interventions: Device: Radiofrequency Ablation System or Microwave Ablation System

INTERVENTIONS:
Device: Multimodal Tumor Thermal Therapy System — All subjects were treated with a multi-modal thermal therapy system (Shanghai MAaGI Medical Technology Co., Ltd.) following a temperature-controlled tumor ablation protocol. Complete ablation of intrahepatic lesions was achieved, resulting in no evidence of disease (NED) within the liver. For lesions that could not be fully ablated in a single session, two treatment sessions were performed to attain intrahepatic NED status.
  Arms: Multimodal Tumor Thermal Therapy
Device: Radiofrequency Ablation System or Microwave Ablation System — All subjects were treated with a radiofrequency ablation system or microwave ablation System. Complete ablation of intrahepatic lesions was achieved, resulting in no evidence of disease (NED) within the liver. For lesions that could not be fully ablated in a single session, two treatment sessions were performed to attain intrahepatic NED status.
  Arms: Single Thermal Ablation

SUMMARY:
Multimodal thermal therapy (MTT), as an initiative integration of cryotherapy and radiofrequency heating, has been applied to treat various solid tumors. The feasibility and safety for MTT in the treatment of malignant liver tumors is well-established. This prospective, multi-center, randomized controlled clinical study aimed to explore the ablation-induced immune activating response of MTT in the treatment of malignant liver tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years.
2. Clinical diagnosis or pathologic of hepatocellular carcinoma (HCC) or metastatic liver cancers.
3. Intrahepatic lesions with a diameter of ≤5cm, and the number of lesions ≤5.
4. Without extrahepatic metastases; for patients with liver metastases, previously underwent radical resection of the primary lesion without local recurrence.
5. Child-Pugh score ≤7 (Class A or B).
6. Performance status 0-1 (Eastern Cooperative Oncology Group classification).
7. Life expectancy of at least 3 months.
8. Patients who have previously undergone surgery, chemotherapy, targeted therapy, ablation, vascular interventional therapy (TACE, D-TACE, HAIC), or immunotherapy, with an interval of ≥3 weeks since the last treatment.
9. The functional level of major organs must meet the following requirements:

(1) Blood Routine: WBC≥3.0×109/L，ANC≥1.5×109/L，PLT≥50×109/L，HGB≥90 g/L. (2) Liver Function: AST ≤5.0×ULN, ALT ≤5.0×ULN, TBIL ≤2.0×ULN. (3) Renal Function: Cr ≤1.5×ULN or CrCl ≥60 mL/min. (4) Coagulation Function: INR ≤1.5; APTT ≤1.5×ULN. (5) HBV-DNA: HBV-DNA ≤2×10³ IU/mL (*Patients with HBV-DNA >2×10³ IU/mL may be enrolled but must receive antiviral therapy.*)

Exclusion Criteria:

1. Diffuse hepatocellular carcinoma (HCC), or with tumor thrombus in the main portal vein to secondary branches or hepatic veins.
2. Severe liver atrophy or excessively large tumor volume requiring ablation of ≥1/3 of the liver volume.
3. Uncorrectable coagulation dysfunction or severe hematologic abnormalities with a high risk of bleeding.
4. Active bacterial infection or fungal infection.
5. Previous or coexisting malignancies.
6. History of solid organ transplant or hepatic encephalopathy.
7. Current enrollment in another clinical trial or prior exposure to experimental therapies.
8. Pregnant or breastfeeding, or preparing to pregnant.
9. Not suitable to participate in clinical trials judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | At 12 months after the ablation procedure on Day 0
  PFS was defined as the time from the first ablation until local tumor progression, any identification of a new (nontarget) lesion/tumor during follow-up, or death due to any cause (whichever occurs first).
Assessment of immune activating response | In 6 months
  The landscape of the peripheral immune response induced by local ablation in patients with malignant liver tumors.

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | At 6 months after the ablation procedure on Day 0
  Refers to the proportion of patients whose tumors shrink to a certain extent and maintain that response for a specified period, including cases of Complete Response (CR) and Partial Response (PR). Tumor objective response is assessed using mRECIST criteria. At baseline, subjects must have measurable tumor lesions. According to the efficacy evaluation criteria, the outcomes are classified as Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD).
Local Control Rate（LCR） | At 6 months after the ablation procedure on Day 0
  LCR is defined as the proportion of patients demonstrating absence of disease progression at the ablated target site according to mRECIST criteria, as evaluated by diagnostic imaging, without evidence of progressive disease (PD) within the prescribed follow-up period.
Overall Survival (OS) | At 36 months after the ablation procedure on Day 0
  OS refers to the time from the date of enrollment to the date of death due to any cause.
Percentage of Participants With Adverse Events (AEs) Within 3 Months Post Ablation | From time of first ablation (Day 0) up to 3 months post ablation
  Percentage of participants with AEs within 3 months post ablation were reported. An AE was an untoward medical occurrence (sign, symptom or disease) in a participant, and which did not necessarily have a causal relationship with the study medical device.

CONTACTS AND LOCATIONS:
Overall Officials: Lichao Xu, M.D, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No